CLINICAL TRIAL: NCT02560766
Title: A Multicenter, Double-Blind, Placebo Controlled, Parallel Group, Efficacy and Safety Evaluation of HORIZANT (Gabapentin Enacarbil Extended-Release Tablets) in Adolescents Aged 13 to 17 Years Old With Moderate-to-Severe Primary RLS
Brief Title: An Efficacy and Safety Evaluation of HORIZANT in Adolescents With Moderate-to-Severe Primary RLS
Acronym: RLS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP109
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: RLS
Keywords: Restless Leg Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HORIZANT 300 mg (Experimental): HORIZANT 300 mg once daily
  Interventions: Drug: HORIZANT 300 mg
- HORIZANT 600 mg (Experimental): HORIZANT 600 mg once daily
  Interventions: Drug: HORIZANT 600 mg
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HORIZANT 300 mg — HORIZANT 300 mg once daily
  Other Names: Gabapentin Enacarbil Extended-Release Tablets
  Arms: HORIZANT 300 mg
Drug: HORIZANT 600 mg — HORIZANT 600 mg once daily
  Other Names: Gabapentin Enacarbil Extended-Release Tablets
  Arms: HORIZANT 600 mg
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
The primary objective of the trial is to evaluate the efficacy of HORIZANT 300 mg and 600 mg, compared to placebo, at 12 weeks of treatment, for the treatment of Restless Legs Syndrome (RLS) in adolescents (13 to 17 years of age) diagnosed with moderate-to-severe primary RLS.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled, 3 arm, parallel group study of HORIZANT in adolescents (13 to 17 years of age) diagnosed with moderate-to-severe primary RLS. Eligible patients enter a 7-day screening period during which safety assessments are performed. Eligible patients are randomized in a 1:1:1 ratio to HORIZANT 300 mg or 600 mg, or matching placebo, followed by a 12-week treatment period. Patients take the study drug once daily at approximately 5 PM with food. Patients will visit the clinical site on 5 or 6 different occasions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adolescent patients, aged 13 to 17 years, diagnosed with RLS based on the IRLSSG consensus criteria (Allen RP 2014) (Appendix 2).
2. Total RLS severity score of 15 or greater on the IRLS rating scale at Visit 1 (screening) and at Visit 2 (baseline) (Appendix 8).
3. RLS symptoms for at least 4 of 7 consecutive evenings/nights during the screening period.
4. Body weight greater than 33.4 kg and a healthy weight using age-based body mass index (BMI) range 5th-95th percentile at screening and baseline.
5. Negative pregnancy test for all females at screening and baseline. Sexually active patients must agree to use 2 medically accepted methods of contraception, 1 of which is a highly effective method (e.g., hormonal or intrauterine device [IUD]) [the second may be a barrier method (e.g., male condom, female condom, diaphragm or cervical cap)], during the course of the study treatment and for 4 weeks after the last dose of study treatment. For patients using hormonal contraceptives as one of the methods, the contraceptive should be stabilized for at least 3 months prior to screening.

   Female patients who normally abstain from sexual activity may be recruited, providing they remain abstinent during the study, or if they become sexually active, they must agree to use 2 effective methods of birth control as described above.
6. Male patients must agree to use a barrier method (male condom, female condom, diaphragm, or cervical cap) with spermicide for at least 30 days prior to dosing and throughout the study, if sexually active. Male patients who normally abstain from sexual activity may be recruited, providing they remain abstinent during the study, or if they become sexually active, they must agree to use a barrier method as described above.
7. Estimated creatinine clearance of at least 60 mL/min (using the Cockcroft-Gault equation) at screening only.
8. Appropriate cognitive and communication skills, as judged by the clinician, needed to complete study assessments.
9. Signed patient and parent Institutional Review Board (IRB)-approved informed consent/assent form (as applicable) before any study-related procedures are performed.
10. Willing and able to follow the study procedures.

Exclusion Criteria:

1. History of a primary sleep disorder other than RLS that may significantly affect the symptoms of RLS.
2. Serum ferritin level < 20 ng/mL at screening.
3. History of allergy, hypersensitivity, or intolerance to HORIZANT or any other gabapentin products (e.g., Neurontin®, Gralise®).
4. Suffering from an isolated periodic limb movement disorder without RLS.
5. Currently meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for substance use disorder, or history thereof, within 12 months before dosing.
6. Current or past history of any significant psychiatric disorder including, but not limited to, depression (treatment with antidepressants), bipolar disorder, or schizophrenia.
7. Diagnosis of ADHD is allowed, provided the patient is not receiving medication(s) known to affect the assessment of RLS.
8. History of suicidal behavior or suicidal ideation as indicated by the C-SSRS, administered at screening, and as per investigator's judgment.
9. Patients with a history of epilepsy, subjects currently prescribed treatments for epilepsy, or subjects with a history of seizure in the last 5 years.
10. Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of gabapentin enacarbil, or, in the Principal Investigator's judgment is considered to be clinically significant and may pose a safety concern, or, could interfere with the accurate assessment of safety or efficacy, or could potentially affect a patient's safety or study outcome.
11. In the judgement of the Principal Investigator, clinically significant, abnormal laboratory result or physical examination finding not resolved by the time of baseline assessments.
12. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody at screening.
13. Uncontrolled hypertension defined as blood pressure (BP) ≥ 95 percentile adjusted for age, height, and sex, according to the tables published by the US Department of Health and Human Services 2005, at screening and before dosing. Appendix 5 contains the tables that can be consulted.
14. Participated in an investigational drug trial within the 4 weeks before dosing or plans to participate in another study at any time during this study.
15. Received an investigational product within 6 months prior to dosing.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
the change on the IRLS rating scale from baseline to Week 12 | 12 weeks
  IRLS rating change
the proportion of patients who are responders, assessed on the CGI-I scale as "much improved" or "very much improved" (CGI-I rating of 1 or 2, respectively) at Week 12 | 12 weeks
  CGI-I scale

SECONDARY OUTCOMES:
IRLS total score, change from baseline to Weeks 4 and 8 | 4, 8 weeks
  IRLS change
CGI-I score at Weeks 4 and 8 | 4, 8 weeks
  CGI-I score
Proportions of patients by sleep parameters collected on the Post-Sleep questionnaire at baseline and Week 12 | Baseline to 12 weeks
  sleep parameters on Post-Sleep questionnaire
Proportions of patients by sleep parameters collected on the ESS-CHAD© total score and change from baseline to Week 12 | Baseline to 12 weeks
  sleep parameters by ESS-CHAD© total score and change
Proportions of patients with AEs, fatal serious adverse events (SAEs), non-fatal SAEs, and discontinuations due to AEs at all post-dose time points; and proportion of patients with neuropsychiatric AEs | 12 weeks
  Adverse event proporations

CONTACTS AND LOCATIONS:
Overall Officials: Steven Caras, MD, Study Director — Xenoport/Arbor Pharmaceuticals, LLC
Locations (12):
- United States (12):
  - Stanford Sleep Medicine Center, Redwood City, California
  - NW FL Clinical Research Group, Gulf Breeze, Florida
  - Orlando Pediatric Pulmonary and Sleep, Winter Park, Florida
  - PANDA Neurology/CIRCA, Atlanta, Georgia
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Pacific Research Network, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Mercy Health - Children's Hospital Pulmonary & Sleep Center, Toledo, Ohio
  - The Sleep Center at the Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - SleepMed of South Carolina; SleepMed, Inc., Columbia, South Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Road Runner Research, San Antonio, Texas